CLINICAL TRIAL: NCT05136716
Title: Long Term Effect of Hyperbaric Oxygen Therapy on Gait and Functional Balance Skills in Cerebral Palsy
Brief Title: Effect of Hyperbaric Oxygen Therapy on Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Mohamed A. Abdel Ghafar, Associate Professor, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyperbaric and Cerebral Palsy
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Cerebral Palsy; Hyperbaric Oxygen Therapy
Keywords: Spastic cerebral palsy; Hyperbaric oxygen therapy; Functional Balance; Gait parameters
MeSH Terms: conditions — Cerebral Palsy | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Children in this group received traditional physical therapy
  Interventions: Other: Traditional Physical Therapy
- Study (Experimental): Children in this group received the same traditional physical therapy plus hyperbaric oxygen therapy
  Interventions: Device: Hyperbaric oxygen therapy

INTERVENTIONS:
Other: Traditional Physical Therapy — Stretching for tight muscles, strengthening for weak muscles, postural reactions training, proprioceptive training, and walking training were all part of the neurodevelopmental treatment plan.
  Arms: Control
Device: Hyperbaric oxygen therapy — HBO2 therapy at a pressure of 1.7 atm For 60 minutes, participants breathed 100% O2.
  Arms: Study

SUMMARY:
Abnormal gait is a common issue in children with CP. As a result of motor weakness and a lack of voluntary motor control. Furthermore, gait in children with cerebral palsy is characterized by a slower walking speed, a shorter stride length, and more time spent in double support. Deficits in postural control constitute a major limitation to the motor development in children with CP. The performance of static and dynamic tasks, such as sitting, standing, and walking, is limited in these children due to postural instability. Postural control deficits in CP are caused by altered sensory processing, motor impairment, and biomechanical alignment, which result in altered neuromuscular responses.

HBO2 therapeutic benefits in CP are attributed to an increase in dissolved oxygen in plasma and tissue, which aids tissue regeneration, So, the purpose of this study was to investigate the long-term effects of hyperbaric oxygen therapy on spatiotemporal gait parameters and functional balance skills in children with CP.

DETAILED DESCRIPTION:
This was a randomized clinical trial. Thirty-nine children with spastic cerebral palsy with ages ranging from 5 to 10 years referred from local pediatric rehabilitation centers participated in this study. All children were classified randomly using sealed envelopes into two groups (Control and Study groups). The children in the control group received traditional physical therapy and the study group received the same traditional physical therapy in addition to hyperbaric oxygen therapy. Written informed consent from the child's legal guardian was obtained. The study was authorized by the Ethics Committee for Research at Cairo University in accordance with the ethical standards of the Declaration of Helsinki. PBS was used to assess functional balance and GAITRite was used to assess spatiotemporal gait parameters. Measurements of functional balance and spatiotemporal gait parameters were taken three times: at the start of the intervention, eight weeks later, and six months after cessation of HPO2 therapy to assess the long-term effect.

ELIGIBILITY:
Inclusion Criteria:

* medically free by their doctor.
* being able to tolerate a hyperbaric oxygen hood.
* being able to blow through a straw, or swallow on command.
* having spasticity ranging from 1 to 1+ on the Modified Ashworth Scale
* level I or II on the Gross Motor Function Classification System (GMFCS).
* being capable of understanding and following instructions

Exclusion Criteria:

* Previous HBO treatments.
* botulinum toxin A treatments.
* thoracic surgery within 6 months.
* major changes to spasticity medications within 3 months.
* unstable epilepsy.
* pulmonary dysfunction.
* cardiovascular disease

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-13 (Actual)

PRIMARY OUTCOMES:
Velocity (cm/s) | 6 months
  Change of the velocity was measured using GAITRite System
Stride Length (cm) | 6 months
  Change of the stride length was measured using GAITRite System
Double leg support (% of gait cycle) | 6 months
  Change of the double leg support was measured using GAITRite System
Functional Balance skills (score) | 6 months
  Change of balance scores was measured using pediatric balance scale. PBS collect scores for the 14 tasks assessed. The tasks are scored on a five-point scale (0, 1, 2, 3 or 4), with zero denoting an inability to perform the activity without assistance and four denoting the ability to perform the task with complete independence. Score range from 0 to 56, with higher scores indicating better postural control

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. AbdelGhafar, Ph.D, Principal Investigator — Batterjee Medical College
Locations (1):
- Batterjee Medical College, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No